CLINICAL TRIAL: NCT01669473
Title: A Primary Care, EHR- Based Strategy to Promote Safe and Appropriate Drug Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Bruce Lambert, Director, Center for Communication and Health, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1U19HS021093-01 (AHRQ)
Record Dates: First submitted 2012-08-03; First posted 2012-08-21 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus Type I; Diabetes Mellitus Type II
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm (Experimental): EHR Based Strategy to promote Safe and Appropriate Drug Use
  Patients randomized to the intervention arm will be given (3) print tools to assist in safe and appropriate medication use. These include a Medreview, Medsheet,and Medlist.
  Interventions: Other: EHR Based Strategy to promote Safe and Appropriate Drug Use
- Standard Care Arm (No Intervention): The control group will receive regular standard care at the Clinic. They will not receive any print tools.

INTERVENTIONS:
Other: EHR Based Strategy to promote Safe and Appropriate Drug Use — The printed tools presented in the intervention include:
  1. Medication Review: a consolidated list of the medications a patient is currently taking.
  2. Medication Sheet: a medication information sheet, including simplified prescription instructions, for each medication that a patient is newly prescribed.
  3. Medication List: a table that lists all medications taken by the patient and provides an orientation on how to best organize and simplify their medication regimen
  Arms: Intervention Arm

SUMMARY:
This study seeks to evaluate a low-literacy strategy in a primary health care setting for promoting safe and effective prescription medication use among English and Spanish-speaking patients with diabetes.

The investigators hypothesize that in comparison with patients receiving standard care, the patients that received the Electronic Health Record (EHR) strategy will 1) demonstrate better understanding of how to safely dose out their medication regimen; 2) have fewer discrepancies in their medication lists; 3) take their medication regimen more efficiently; 4) have greater adherence to their medication regimen.

DETAILED DESCRIPTION:
The strategy takes advantage of health information technology to assist patients with Medication Therapy Management (MTM) tasks, intervening with a set of low-literacy MTM printed tools triggered by the Electronic Health Record (EHR) in a primary health care clinic. Patients at the University of Illinois at Chicago (UIC) Medicine Clinic who are randomized to the intervention arm will be given three printed tools, one when they check in to the clinic and the other two when they check out. The Electronic Health Record (EHR) triggers the printing of these tools, and the receptionist hands them to the patient. Patients receive either English or Spanish language materials depending on the preference determined in the screening process and stored in their EHR.

Specific Aims

1. Refine and Field Test an EHR strategy for generating and distributing low literacy prescription information for English and Spanish-speaking patients
2. Assess the process of the EHR intervention and its fidelity for providing prescription information for patients at the point of prescribing and dispensing medications.
3. Evaluate the effectiveness of the EHR strategy to improve medication understanding, reconciliation, regimen consolidation, and adherence compared to standard care.

In addition, we will be powered to also investigate our strategy's impact on intermediary clinical outcomes including systolic blood pressure, HbA1c, and LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* 18-years old or older;
* have a diagnosis of diabetes mellitus either by ICD-billing codes or indicative medications;
* are prescribed at least (3) chronic condition medications according to the EHR medication list;
* are English or Spanish-speaking;
* have no imminent intention to move or change clinics within the next year;
* score 4 or higher on the six-question screener based on the Mini-Mental Status Exam;
* are primarily responsible for administering their own medications;
* prescribed a new chronic condition medication (including refills, and change in titrations) during their clinic visit and day.

Exclusion Criteria:

* under age of 18 years-old;
* does not speak English or Spanish;
* dependent on assistance for medication administration;
* scored less than 4 on the six-question screener;
* not prescribed a new medication or changed medication at clinical appointment;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2013-06; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Medication adherence | One month after patients receive intervention materials
  We will determine to what extent presenting low-literacy information about prescription medicines to patients with diabetes affects their adherence to a medication regimen compared to patients under standard care.
  Adherence for each prescription medication will be measured through multiple methodologies.

SECONDARY OUTCOMES:
Clinical outcomes-systolic blood pressure, HbA1, and LDL cholesterol. | Baseline interview and after 6 months
  We will investigate our strategy's impact on intermediary clinical outcomes including systolic blood pressure for patients with hypertension, HbA1 for patients with diabetes, and LDL cholesterol for patients with hyperlipidemia, through chart extraction at pre and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Lambert, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois

REFERENCES:
- [Derived] Przytula K, Bailey SC, Galanter WL, Lambert BL, Shrestha N, Dickens C, Falck S, Wolf MS. A primary care, electronic health record-based strategy to promote safe drug use: study protocol for a randomized controlled trial. Trials. 2015 Jan 27;16:17. doi: 10.1186/s13063-014-0524-x. PMID 25622970